CLINICAL TRIAL: NCT07101627
Title: A Prospective, Multicenter Clinical Study of Hetrombopag in the Prevention of Thrombocytopenia Caused by Lung Cancer Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ren Shengxiang, professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MA-CTIT-II-013
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — hetrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hetrombopag Tablets (Experimental): patients will receive oral administration of hetrombopag, 7.5 mg/day, for 14 days from the first day after the end of chemotherapy in this cycle.
  Interventions: Drug: Hetrombopag Tablets
- Hetrombopag Simulated Tablets (Placebo Comparator): patients in the control group began to orally take hetrombopag simulated tablets 7.5 mg/day for 14 days on the first day after the end of chemotherapy in this cycle.
  Interventions: Drug: Hetrombopag Tablets

INTERVENTIONS:
Drug: Hetrombopag Tablets — Stage 1: After screening and enrollment, patients will receive oral administration of hetrombopag, 7.5 mg/day, for 14 days from the first day after the end of chemotherapy in this cycle.
  Stage 2: Patients who met the inclusion criteria were randomized 1:1 to the experimental group and the control group after enrollment. Patients in the experimental group began to orally take hetrombopag 7.5 mg/day for 14 days on the first day after the end of chemotherapy in this cycle; patients in the control group began to orally take hetrombopag simulated tablets 7.5 mg/day for 14 days on the first day after the end of chemotherapy in this cycle. Randomization was stratified by concomitant immunotherapy (yes versus no) and chemotherapy with gemcitabine plus platinum (yes versus no).

SUMMARY:
To evaluate the efficacy and safety of Hetrombopag in secondary prevention of thrombocytopenia caused by lung cancer treatment

DETAILED DESCRIPTION:
The study was divided into 2 study periods, Stage 1 was a prospective, single-arm study design and Stage 2 was a prospective, randomized, double-blind, placebo-controlled study design. According to the results of Phase 1 study, Phase 2 study design and sample size were confirmed.

Stage 1: After screening and enrollment, patients will receive oral administration of hetrombopag, 7.5 mg/day, for 14 days from the first day after the end of chemotherapy in this cycle.

Stage 2: Patients who met the inclusion criteria were randomized 1:1 to the experimental group and the control group after enrollment. Patients in the experimental group began to orally take hetrombopag 7.5 mg/day for 14 days on the first day after the end of chemotherapy in this cycle; patients in the control group began to orally take hetrombopag simulated tablets 7.5 mg/day for 14 days on the first day after the end of chemotherapy in this cycle. Randomization was stratified by concomitant immunotherapy (yes versus no) and chemotherapy with gemcitabine plus platinum (yes versus no).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be enrolled in the study：

  1. Age ≥ 18 years, gender is not limited.
  2. Patients with histopathologically confirmed metastatic lung cancer.
  3. Receiving platinum- or gemcitabine-based (21-day chemotherapy cycles) antineoplastic therapy with an anticipated treatment of ≥ 2 cycles.
  4. ECOG PS score 0-2.
  5. Platelet count < 75 × 10^9/L in previous cycle due to same lung cancer treatment regimen.
  6. PLT between 100-200 × 10^9/L prior to enrollment.
  7. Primary organ function normal:

     ① Bone marrow hematopoiesis: ANC ≥ 1.5×10^9/L; hemoglobin ≥ 8 g/dL;

     ② Liver and kidney function: total bilirubin ≤ 1.5 ULN; ALT, AST ≤ 2.5 ULN; if liver metastasis is present, ALT, AST ≤ 5 ULN; serum creatinine ≤ 1.5 ULN or creatinine clearance > 60 mL/min (Cockcroft-Gault);

     ③ Coagulation function: activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5 ULN
  8. Expected survival ≥ 3 months.
  9. Female subjects of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose and not breastfeeding and must agree to use effective contraception during the trial and for 7 days after the last dose of study drug; male subjects with partners of childbearing potential should be surgically sterilized or agree to use effective contraception during the trial and for 7 days after the last dose of study drug and are not allowed to donate sperm during the study.
  10. Voluntarily join this study, sign informed consent form, have good compliance and are willing to cooperate in follow-up.

Exclusion Criteria:

* Subjects will not enter this study if they have any of the following characteristics or conditions:

  1. Pregnant or lactating women.
  2. Inability to understand the investigational nature of the study or lack of informed consent.
  3. Associated hematopoietic disorders, including but not limited to leukemia, primary immune thrombocytopenia, myeloproliferative disorders, multiple myeloma, and myelodysplastic syndrome.
  4. Other diseases causing thrombocytopenia other than thrombocytopenia caused by anti-tumor therapy (CTIT) within 6 months before screening, including but not limited to chronic liver disease, hypersplenism and infection.
  5. Presence of active uncontrolled infection.
  6. Tumor bone marrow invasion or bone marrow metastasis.
  7. Any arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism) within 6 months prior to Screening, or clinical symptoms and history suggestive of thrombophilia.
  8. Cardiac disorders, including Grade 3/4 congestive heart failure, cardiac arrhythmia or myocardial infarction requiring medication, or cardiac arrhythmia known to increase the risk of thrombotic events (eg, atrial fibrillation), or prolongation of the subject 's corrected QT interval (QTc) within 3 months prior to Screening.
  9. Thrombocytopenia not due to antineoplastic therapy.
  10. Known hypersensitivity to TPO.
  11. Patients accompanied by severe bleeding symptoms or with clear clinical manifestations of bleeding tendency, such as gastrointestinal tract or cerebral hemorrhage.
  12. Concurrent use of other drugs that may affect platelet count (traditional Chinese medicine, proplatelet, antiplatelet, etc.)
  13. Other conditions not suitable for inclusion in the study judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 and Higher Thrombocytopenia | One cycle of treatment(21 days)
  Incidence of platelet count ≤ 50 × 10^9/L

SECONDARY OUTCOMES:
Incidence of Grade 2 and Higher Thrombocytopenia | One cycle of treatment(21 days)
  Incidence of platelet count ≤ 75 × 10^9/L
Platelet count nadir | One cycle of treatment(21 days)
  Platelet count nadir
The time it takes for PLT to recover from the lowest value to ≥100×10^9/L | One cycle of treatment(21 days)
  The time it takes for PLT to recover from the lowest value to ≥100×10^9/L
Duration of Grade 3 or Higher Thrombocytopenia | One cycle of treatment(21 days)
  Duration of platelet count ≤ 50 × 10^9/L
Platelet count on the day before the next cycle of chemotherapy | The day before the next cycle of chemotherapy
  Platelet count on the day before the next cycle of chemotherapy
Proportion of patients with a delay, dose reduction, suspension, or regimen modification of their next cycle of antineoplastic therapy due to thrombocytopenia | One cycle of treatment(21 days)
  Proportion of patients with a delay, dose reduction, suspension, or regimen modification of their next cycle of antineoplastic therapy due to thrombocytopenia
Proportion of Salvage Patients | One cycle of treatment(21 days)
  Proportion of Salvage(Platelet transfusion, interleukin-11, recombinant human thrombopoietin) Patients
Safety(The occurrence of any AEs ) | One cycle of treatment(21 days)
  Adverse events (evaluated using NCI CTCAE Version 5.0), laboratory tests, vital signs, electrocardiograms, and physical examinations, as well as the incidence and severity of bleeding events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai, China, Shanghai, Shanghai Municipality